CLINICAL TRIAL: NCT02313337
Title: The Comparison of Different Administration Routes of Pediatric Premedication-Single Center,Randomized，Controlled Trial
Brief Title: The Comparison of Different Administration Routes of Pediatric Premedication
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: administration route
Record Dates: First submitted 2014-11-27; First posted 2014-12-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-11

CONDITIONS: Anesthesia
Keywords: Administration route; Preanesthetic medication; Sedation
MeSH Terms: interventions — Administration, Oral; Injections, Intramuscular; Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Oral administration (Experimental): -Oral administration of a mixture at preoperative 30 minutes : ketamine 3 mg/kg, midazolam 0.5 mg/kg and atropine 0.02 mg/kg, plus 50% glucose solution to 0.5ml /kg.
  Interventions: Other: Oral administration; Drug: Anesthesia induction(midazolam,fentanyl,propofol,atracurium); Procedure: Intubation; Drug: Anesthesia maintenance(midazolam,fentanyl,propofol,atracurium)
- Intramuscular injection (Experimental): -At preoperative 30 minutes intramuscular injection of atropine 0.02 mg/kg, 5 minutes before entering the operation room, intramuscular injection of ketamine 5 mg/kg.
  Interventions: Other: Intramuscular injection; Drug: Anesthesia induction(midazolam,fentanyl,propofol,atracurium); Procedure: Intubation; Drug: Anesthesia maintenance(midazolam,fentanyl,propofol,atracurium)
- Rectal perfusion (Experimental): -At preoperative 30 minutes rectal infusion of midazolam 0.5mg/kg
  Interventions: Other: Rectal perfusion; Drug: Anesthesia induction(midazolam,fentanyl,propofol,atracurium); Procedure: Intubation; Drug: Anesthesia maintenance(midazolam,fentanyl,propofol,atracurium)
- Dripping nose (Experimental): -At preoperative 30 minutes dripping nose of Imidazole valium 0.2 mg/kg
  Interventions: Other: Dripping nose; Drug: Anesthesia induction(midazolam,fentanyl,propofol,atracurium); Procedure: Intubation; Drug: Anesthesia maintenance(midazolam,fentanyl,propofol,atracurium)

INTERVENTIONS:
Other: Oral administration — Premedicate--Oral administration of a mixture at preoperative 30 minutes: ketamine 3 mg/kg, midazolam 0.5 mg/kg and atropine 0.02 mg/kg, plus 50% glucose solution to 0.5ml /kg.
  Arms: Oral administration
Other: Intramuscular injection — Premedicate--At preoperative 30 minutes intramuscular injection of atropine 0.02 mg/kg, 5 minutes before entering the operation room, intramuscular injection of ketamine 5 mg/kg.
  Arms: Intramuscular injection
Other: Rectal perfusion — Premedicate--At preoperative 30 minutes rectal infusion of midazolam 0.5mg/kg
  Arms: Rectal perfusion
Other: Dripping nose — Premedicate--At preoperative 30 minutes dripping nose of Imidazole valium 0.2 mg/kg
  Arms: Dripping nose
Drug: Anesthesia induction(midazolam,fentanyl,propofol,atracurium) — After entering the operation room ,all cases intravenous midazolam 0.05 mg/kg, fentanyl 3μg/kg, closed-loop target controlled infusion propofol and atracurium .
Procedure: Intubation — Intubation when the trachea-oesophageal fistula（TOF） value fell 15%, BIS value dropped to 40.
Drug: Anesthesia maintenance(midazolam,fentanyl,propofol,atracurium) — All cases intravenous midazolam 0.05 mg/kg, fentanyl 3μg/kg, closed-loop target controlled infusion propofol and atracurium .

SUMMARY:
The study purpose is to compare the effect of different Administration Routes of Pediatric Premedication (including oral administration, intramuscular injection, rectal perfusion, intranasal).

DETAILED DESCRIPTION:
In this study, 80 cases of surgical or otolaryngology children undergoing elective surgery were divided into four groups：oral administration group, intramuscular group, rectal infusion group, intranasal group depending on the route of administration before anesthesia. By observing the difference of sedative effects, postoperative recovery, and postoperative psychological behavior among the four groups,compare the effect of four pre-anesthetic administration routes.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent of children's parents;
* Children patient in pediatric surgery and E.N.T. department;
* surgery time 1 ~ 3 hours;
* Aged between 1 and 7 years old;
* American Society of Anesthesiologists (ASA)classification:class I~II;

Exclusion Criteria:

* With cardiovascular and respiratory complications;
* A history of the endocrine system;
* A long history of application of sedative drugs;
* Water and electrolyte balance disorder preoperatively;
* Liver and kidney dysfunction;
* Nervous system dysfunction;
* High gastrointestinal obstruction;
* Tracheoesophageal fistula, trachea foreign body, hiatal hernia, dysphagia;
* Lung infection, atelectasis;
* Congenital heart disease(CHD);
* Severe malnutrition;
* Traumatic or ischemia anoxic encephalopathy, high cranial pressure;
* Anesthesia and surgery was conducted in 3 days;

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Sedation Score | Try to break away from family membersan，an expected average of 3 min；Successfully break away from the family members and accept the face mask and venipuncture，an expected average of 5 min

SECONDARY OUTCOMES:
Hemodynamic and anesthetic depth monitoring (Heart rate, blood pressure, pulse oxygen saturation, bispectral index(BIS) | From premedication to 10 min after extubation up to 4 hours
  Heart rate, blood pressure, pulse oxygen saturation, bispectral index(BIS)
Stress index monitoring (The concentration of Plasma cortisol and blood sugar) | From anesthesia induction to 10 min after the start of surgery up to 30 min
  The concentration of Plasma cortisol and blood sugar
Postoperation recovery assess (Wake up agitation score (PAED)、Steward score 、Postoperative recovery score) | 10 min after extubation
  Wake up agitation score (PAED)、Steward score 、Postoperative recovery score
Postoperative behavior assessment (Postoperative behavior scale (PHBQ) | 1 day after the operation，7 day after the operation
  Postoperative behavior scale (PHBQ)

CONTACTS AND LOCATIONS:
Overall Officials: NIU XIAOLI, Principal Investigator — The second affiliated hospital of xi 'an jiaotong university

REFERENCES:
- [Background] Haas U, Motsch J, Schreckenberger R, Bardenheuer HJ, Martin E. [Premedication and preoperative fasting in pediatric anesthesia. Results of a survey]. Anaesthesist. 1998 Oct;47(10):838-43. doi: 10.1007/s001010050633. German. PMID 9830555
- [Background] Kain ZN, Mayes LC, Bell C, Weisman S, Hofstadter MB, Rimar S. Premedication in the United States: a status report. Anesth Analg. 1997 Feb;84(2):427-32. doi: 10.1097/00000539-199702000-00035. PMID 9024042